CLINICAL TRIAL: NCT06084156
Title: A Phase I Clinical Study to Evaluate the Drug-Drug Interaction Between HSK7653 and Metformin in Healthy Subjects
Brief Title: A Study to Evaluate the DDI of HSK7653 With Metformin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSK7653-102
Record Dates: First submitted 2023-09-24; First posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-09

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HSK7653 and Metformin (Experimental)
  Interventions: Drug: HSK7653; Drug: Metformin

INTERVENTIONS:
Drug: HSK7653 — Part 1: Day 1 to Day 4, not take; Part 2: Day 6 - Take HSK7653 35 mg; HSK7653 25 mg on day 13, day 20, day 27, and day 34; Part 3: Day 41 - Take HSK7653 25 mg
Drug: Metformin — Part 1: Day 1 to Day 4, 1000mg BID; Part 2: Not take; Part 3: Day 38- day 47, 1000mg BID

SUMMARY:
This is a Phase 1, single center, open-label, single arm, drug-drug interaction study of HSK7653 and metformin in Healthy Subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and Age ≤60 years
* BMI ≥18 and BMI ≤ 28 kg/m2 (Body Mass Index)
* Able to understand the procedures of the study, and provide written informed consent and willing to comply with the study protocol procedures.

Exclusion Criteria:

* Any finding of the medical examination (physical examination, laboratory examination, 12-ECG, abdominal B-ultrasonography, etc) deviating from normal and of clinical relevance during screening;
* Fasting blood glucose <3.9mmol/L or ≥6.1mmol/L;
* Has a condition affecting the absorption, distribution, metabolism, and excretion of the drug;
* Has a positive result on screening for serum hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCVAb), Treponema pallidum antibody (TP-Ab) or human immunodeficiency virus (HIV);
* Treatment with an investigational drug within 3 months;
* Other protocol-defined exclusion criteria.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2019-08-10 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2019-12-09 (Actual)

PRIMARY OUTCOMES:
The primary pharmacokinetics parameter of Cmax To assess the potential pharmacokinetic interaction between HSK7653 and metformin in health subjects. | Day4, day 27 and day 41
The primary pharmacokinetics parameter of AUC To assess the potential pharmacokinetic interaction between HSK7653 and metformin in health subjects. | Day4, day 27 and day 41

SECONDARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (TEAEs) | First dose of study drug up to 62 days after last dose of study drug
Pharmacodynamic responses of glucose, insulin and C-peptide will be evaluated | Day 41

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No